CLINICAL TRIAL: NCT02756221
Title: The Effect of Probiotic Supplementation on the Incidence of Gastrointestinal (GI) Tract and Upper Respiratory System Symptoms and the Endurance Exercise Performance in Masters Runners and Elite Cyclists
Brief Title: Probiotic Supplementation and Endurance Performance in Cyclists and Masters Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Principal Investigator, Itzik Weinstein, Head Exercise Physiology Laboratory, Tel Hai College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Exercise Testing
Record Dates: First submitted 2016-04-11; First posted 2016-04-29 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Viral Upper Respiratory Tract Infection; Gastroenteritis
Keywords: symptoms
MeSH Terms: conditions — Gastroenteritis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Experimental): Probiotics capsules, one capsule daily for 90 days.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Starch capsules, one capsule daily for 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — One capsule per day for 90 days. Containing 8 x 109 CFU of bacteria /capsule Lactobacillus heleveticus Lafti L10 Bifidobacterium animalis ssp lactis Lafti B94 Enterococcus faecium Rosell-26 Bifidobacterium longum RO175 Bacillus subtills Rosell-179 Inactive ingredients: potato starch, magnesium stearate, ascorbic acid White vegetable capsule size 1
  Other Names: Taam Teva Digestion Caps
  Arms: Probiotics
Other: Placebo — Placebo capsules identical in shape and color to the probiotics capsules, one capsule per day for 90 days
  Arms: Placebo

SUMMARY:
The study will evaluate the change in gastrointestinal (GI) flora following probiotic supplementation, and expected to lead to an increase in the intestinal epithelial integrity and to improvement in its health. Concurrently with the reduction in the amount of toxins in the GI tract following an intensive exercise, a lower incidence of symptoms of discomfort will improve the quality of the training sessions which will be exhibited by an improvement in endurance capacity and in physiological responses to rigorous exercise. Half of the participants will receive probiotic supplement while the other half will receive a placebo.

DETAILED DESCRIPTION:
Masters runners and professional competitive cyclists will be recruited, as follows: 30 young road cyclists ages 18-39 years, 60 masters runners ages 40-60 years

Sample Size: 90 subjects will be recruited, following the first set of tests and experiments will randomly be divided into two matched groups experimental and experimental groups. The rational for sample size calculation is based on detecting a defined effect size with 5% statistical significance and 80% power. Effect size reflects the difference in the treatment effect between the groups will be calculated as the difference in measurement values between the experimental (probiotics) and control (placebo) groups divided by the standard deviation. Cyclists' cohort will include 34 subjects which will demonstrate effect size of 1.0. Masters runners' cohort will include 60 subjects which will demonstrate effect size of 0.75.

Study design: A random double-blind prospective study

Recruitment of participants will be executed by study staff which will also serve as trainers of cycling and running groups in Israel's Upper Galilee area.

Subsequently to signing on an informed consent form with one of the study physicians, participants will complete the following procedures:

* A series of preliminary tests (Anthropometry, Maximal Oxygen Consumption, Endurance tests) will be conducted by one of the study physicians from Ziv Medical Center in Zefat
* Food Frequency Questionnaires (FFQ ) and frequency of GI symptoms will be completed electronically with Qualtrics (Qualtrics LLC, Provo, UT, USA)
* Blood samples (approximately 10 ml of venous blood) for quantifying immune factors (inflammation) will be collected at Ziv Medical Center or at Tel Hai Academic College and will be sent to the molecular microbiology and biotechnology laboratory in Tel Aviv University.
* Stool samples for testing the genetic expression of the microbiome composition. The tests will be delivered to the study staff at Tel Hai University and after freezing them, they will be sent together in dry ice to the molecular microbiology and biotechnology laboratory in Tel Aviv University
* Tests for evaluating aerobic endurance (Lactate Threshold - cyclists, running economy or time to fatigue - runners) will be conducted at the exercise physiology laboratory in Tel Hai College.

After the completion of tests, participants will randomly be divided to 2 matched groups according to the level of physical fitness, and age in a double-blind design. The experimental (E) group will be given probiotic supplement in capsule form whereas the control (C) group will be given placebo capsules identical in size and color to the probiotic ones.

The participants will consume the supplement / placebo capsules during a period of 90 days after which they will return for an additional visit in which they will re-complete questionnaires and will undergo identical tests and procedures which they had completed during their first visit (before the assignment into groups).

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* at least 3 years of national-level experience, including participation in competitions
* suffer from one or more of the following symptoms: nausea, vomiting, belching, heartburn and chest pain, bloating, cramps, side pain, urge to empty bowels and diarrhea during training and competitions

Exclusion Criteria:

* Diagnosis of gastrointestinal diseases
* Diagnosis of heart diseases
* Use of Probiotics during the 3 months' period prior to the study
* Use of Antibiotics during the 3 months' period prior to the study
* A radical surgery in the digestive system during the year prior to the

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2max) | 90 days
  Maximal oxygen consumption (VO2max, l/min, or ml/min/kg) is expected to rise following 2 months of supplementation
Ventilatory threshold (VTH) | 90 days
  Ventilatory threshold (VTH), determined during a graded exercise test which measures maximal oxygen consumption (VO2max), and is the deflection point of CO2 production vs VO2 and is expressed as the running speed (km/h) at which it is occurs, and also as percentage of VO2max. Following 3 months of supplementation a right shift in the VTH curve is expected indicating an improved aerobic endurance, meaning that it is occurring at a higher running velocity (km/h)
Running economy | 90 days
  Running economy calculated from the slope of oxygen consumption (VO2) vs 3-4 submaximal running velocities (km/h) is expected to improve, the lower the slope (Liter Oxygen/km/hour) the better the running economy
Time to Fatigue | 90 days
  Time to fatigue (minute; seconds) calculated as at exercise intensity of 85-88% of VO2max is expected to rise, increased time to fatigue indicates improved aerobic endurance

CONTACTS AND LOCATIONS:
Overall Officials: Ron Golan, MD, Principal Investigator — Ziv Medical Center, Zefat, Israel
Locations (1):
- Exercise Physiology Laboratory, Tel H̱ay, Israel

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual subjects data for all outcome measures will be made available within 12 months of study completion

REFERENCES:
- [Result] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Result] Coyle EF. Integration of the physiological factors determining endurance performance ability. Exerc Sport Sci Rev. 1995;23:25-63. PMID 7556353
- [Derived] Schreiber C, Tamir S, Golan R, Weinstein A, Weinstein Y. The effect of probiotic supplementation on performance, inflammatory markers and gastro-intestinal symptoms in elite road cyclists. J Int Soc Sports Nutr. 2021 May 17;18(1):36. doi: 10.1186/s12970-021-00432-6. PMID 34001168